CLINICAL TRIAL: NCT01125722
Title: Pilot Clinical Trial to Study the Effectiveness of a Four-week Exposure to a Transcutaneous, High-frequency, Amplitude-modulated, Non-invasive Neurostimulation Device on Urgency (Urinary) Incontinence in Subjects With Idiopathic Overactive Bladder (OAB)
Brief Title: Clinical Trial to Study a Non-invasive Neurostimulation Device on Urgency (Urinary) Incontinence Overactive Bladder (OAB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Collaborators: Novella Clinical (Other); Data & Inference, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-10-0001
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Overactive Bladder
Keywords: Urinary Incontinence; Overactive Bladder; Frequency; Urgency
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigator Placement Group (Active Comparator)
  Interventions: Device: Non-invasive neurostimulation device
- Subject Placement Group (Active Comparator)
  Interventions: Device: Non-invasive neurostimulation device

INTERVENTIONS:
Device: Non-invasive neurostimulation device — Active electrode patches are worn for 4 weeks, one per week, during the treatment phase of the study. The patch is placed by the investigator.
  Arms: Investigator Placement Group
Device: Non-invasive neurostimulation device — Active electrode patches are worn for 4 weeks, one per week, during the treatment phase of the study. The patch is placed by the subject.
  Arms: Subject Placement Group

SUMMARY:
The purpose of this study is to determine whether the non-invasive neurostimulation patch is effective in the treatment of urgency, frequency and urge (urinary) incontinence.

DETAILED DESCRIPTION:
While the precise cause of OAB symptoms (urge, frequency, incontinence) is not clear, most physicians and researchers accept the theory that a problem in the communication between the central nervous system and the bladder is a factor.

Research has shown that a process called neuromodulation of the nerves controlling the bladder can overcome this communication problem. In patients who have symptoms caused by the communication problem, neuromodulation has been clinically proven to eliminate or significantly reduce those symptoms. While neuromodulation has been previously achieved by implanting an electrode near the sacral nerve in the spine, the new concept under investigation within this protocol is believed to achieve a similar effect from adhesive electrodes placed on the skin over spinal nerves in the lower back.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy the following criteria in order to be enrolled in the study:

* Males and Females, at least 18 years of age
* Documented symptoms of idiopathic overactive bladder for at least 6 months
* Failure on primary OAB treatment, such as behavior modification or fluid/diet management, AND at least one (1) anti-cholinergic drug
* An average of one (1) or more urgency (urinary) incontinence episodes per 24-hours, confirmed by the 3-day baseline voiding diary, with a maximum of 12 urgency (urinary) incontinence episodes per 24-hours
* An average of eight (8) or more voids per 24-hours, confirmed by the 3-day baseline voiding diary
* Demonstrated ability to adequately complete the 3-day baseline voiding diary
* Willing and capable of understanding and complying with all requirements of the protocol
* Signed Informed Consent to participate in the study after full discussion of the research nature of the treatment and its risks and benefits.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

* Urinary retention
* Clinically significant bladder outlet obstruction
* Morbidly obese, defined as having BMI > 40 kg/m2
* Stress predominant mixed urinary incontinence
* Neurological disease affecting urinary bladder function, including but not limited to Parkinson's disease, multiple sclerosis, stroke, spinal cord injury.
* History of epilepsy
* Pelvic surgery (such as sub-urethral sling, pelvic floor repair) within the past 6 months
* Intravesical or urethral sphincter Botulinum Toxin Type A injections within the past 12 months
* Failure of previous neuromodulation therapy for overactive bladder
* Percutaneous Tibial Nerve Stimulation (PTNS) therapy for overactive bladder within the past 6 months
* Any clinically significant congenital or acquired disorder of the urogenital tract (including denovo OAB following sub-urethral sling)
* Vaginal prolapse greater than Stage II in the anterior compartment of the vagina using International Continence Society (ICS) Pelvic Organ Prolapse Quantification (POPQ) criteria.
* Prior peri-urethral or transurethral bulking agent injections for bladder problems within the past 12 months.
* History of pelvic radiation therapy
* Any skin conditions affecting treatment or assessment of the treatment sites
* History of lower back surgery or injury that could impact placement of the patch, or where underlying scar tissue or nerve damage may impact treatment.
* Unable to operate the device remote control.
* Lacking dexterity to properly utilize the components of the device system.
* Presence of an implanted electro-medical device (e.g. pacemaker, defibrillator, InterStim®, etc.),
* Any metallic implant in the back.
* Pregnant, nursing, suspected to be pregnant (by urine pregnancy method), or plans to become pregnant during the course of the study.
* History of dementia or Alzheimer's disease.
* Known latex allergies
* Uncontrolled diabetes and/or diabetes with peripheral neuropathy.
* Transurethral instrumentation within the preceding month.
* Scheduled for any of the following during the course of the study: Magnetic Resonance Imaging (MRI), Positron Emission Tomography (PET), X-ray, Ultrasound, or Radiotherapy (targeting full body or back region)
* Recurrent Urinary Tract Infections (>3 UTI's in the past year)
* Clean catch Urinalysis results >10wbc/hpf
* History of or current lower tract genitourinary malignancies
* Any clinically significant systemic disease or condition that in the opinion of the Investigator would make the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwani Monga, BM BS, MRCOG, Principal Investigator — Princess Anne Hospital, Southampton, UK
Locations (11):
- United States (9):
  - Medical Faculty Associates, The George Washington University, Washington D.C., District of Columbia
  - William Beaumont Hospital - Department of Urology, Royal Oak, Michigan
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Delaware Valley Urology, LLC, Mount Laurel, New Jersey
  - McKay Urology, Charlotte, North Carolina
  - Alliance Urology Specialists, P.A., Greensboro, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Wheaton Franciscan Medical Group, Milwaukee Urogynecology, Wauwatosa, Wisconsin
- Danderyd University Hospital, Stockholm, Sweden
- Princess Anne Hospital, Southampton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigator Placement Group: Nerve stimulation patch is placed by the investigator at Weeks 1 through 4.
- Subject Placement Group: Nerve stimulation patch is placed by the investigator at Week 1 and then by the subjects at Weeks 2 through 4.
Period: Overall Study
Arm/Group | Investigator Placement Group | Subject Placement Group
Started | 37 | 37
Completed | 34 | 36
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigator Placement Group | Subject Placement Group | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 18 | 43
  >=65 years | 12 | 19 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.6) | 62.1 (14.6) | 60.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 25 | 28 | 53
  United Kingdom | 5 | 3 | 8
  Sweden | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Urgency Incontinence Episodes
Description: Mean urgency incontinence episodes (or urinary leaks) over 24 hours is based on a 3-day diary maintained by the subject. Urgency incontinence is when a subject has urinary leakage, i.e., uncontrolled release of fluid prior to making it to the bathroom. The number of leaks over 3 days was recorded for each subject at baseline and again at Week 4. The 3-day average at each time point was used as the mean over 24 hours and the change from baseline to Week 4 was calculated for each subject.
Time Frame: From baseline to Week 4 of active treatment
Population: Modified Intent-to-Treat Set (Full Analysis Set) - defined as all eligible subjects who were randomized to one of the two treatment arms and received some treatment.
Measure: Mean (Standard Deviation); unit: number of incontinence episodes/24 hours
Arm/Group | Investigator Placement Group | Subject Placement Group
Number analyzed (Participants) | 32 | 37
number of incontinence episodes/24 hours | -2.5 (3.05) | -2.5 (2.98)

2. Secondary Outcome: Change in Mean Daily Voiding Frequency
Description: Mean daily voiding frequency over 24 hours is based on a 3-day diary maintained by the subject. Voiding frequency is defined as the number of times a subject urinates. The number of voids over 3 days was recorded for each subject at baseline and again at Week 4. The 3-day average at each time point was used as the mean over 24 hours and the change from baseline to Week 4 was calculated for each subject.
Time Frame: From baseline to Week 4 of active treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of voids per 24 hours
Arm/Group | Investigator Placement Group | Subject Placement Group
Number analyzed (Participants) | 32 | 37
number of voids per 24 hours | -1.8 (2.13) | -1.6 (2.92)

3. Secondary Outcome: Change in Mean Volume Per Void
Description: Mean volume per void (or amount of urine per urination) over 24 hours is based on a 3-day diary maintained by the subject. The volume of void (in milliliters) over 3 days was recorded for each subject at baseline and again at Week 4. The 3-day average at each time point was used as the mean over 24 hours and the change from baseline to Week 4 was calculated for each subject.
Time Frame: From Baseline to Week 4 of active treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Investigator Placement Group | Subject Placement Group
Number analyzed (Participants) | 32 | 37
mL | 5.3 (26.37) | 10.5 (57.01)

4. Secondary Outcome: Change in Mean Urgency Episodes Per Day
Description: Mean urgency episodes per day is based on a 3-day diary maintained by the subject. An urgency episode is identified by the subject as a case where they have a strong urge to urinate, i.e. difficulty controlling the bladder and thus are rushing to the bathroom. The number of urgency episodes over 3 days was recorded for each subject at baseline and again at Week 4. The 3-day average at each time point was used as the mean over 24 hours and the change from baseline to Week 4 was calculated for each subject.
Time Frame: From Baseline to Week 4 of active treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of urgency episodes per 24 hours
Arm/Group | Investigator Placement Group | Subject Placement Group
Number analyzed (Participants) | 32 | 37
number of urgency episodes per 24 hours | -2.1 (2.47) | -2.1 (3.08)

5. Secondary Outcome: Change in Mean Overactive Bladder Symptom Composite Score
Description: The Overactive Bladder Symptom Composite is a composite symptom score of toilet voids, urgency severity and urge urinary incontinence. It combines the Indevus Urgency Severity Scale for capture of urgency severity per toilet void with 24-hour frequency and urinary urge incontinence episodes. A complete reference for this validated measure can be found in teh Journal of Urology, Vol. 173, pgs 1639-1643, May 2005. The scale is specific to the instrument and lower scores represent an improvement in symptoms. The scale is a weighted average of each void a subject has. The weights are assigned as 0=no urgency, 1=mild, 2=moderate, 3=severe. The minimum score is 0, corresponding to no urgency in every void. There is no quantifiable upper limit since the scale is based on the number of voids per day, but there are reasonable upper limits. For example, if a subject had 15 voids in 1 day and all 15 were severe (=3), the Composite Score would be 45. Full details are in the reference above.
Time Frame: From Baseline to Week 4 of active treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Investigator Placement Group | Subject Placement Group
Number analyzed (Participants) | 32 | 37
scores on a scale | -11.7 (16.52) | -11.7 (14.58)

ADVERSE EVENTS:
Arm/Group | Investigator Placement Group | Subject Placement Group
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 16/37 | 14/37
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigator Placement Group (N=37) | Subject Placement Group (N=37)
Skin Reaction (Skin and subcutaneous tissue disorders) | 14 (27) | 12 (22)
Sensory/Peripheral Neurological Effect (Nervous system disorders) | 3 (4) | 3 (3)
Urinary Tract Reactions (Renal and urinary disorders) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No